CLINICAL TRIAL: NCT02158741
Title: A Client-Driven Intervention to Support Self-Management Among Community-Living Older Adults With Type 2 Diabetes and Multiple Chronic Conditions
Brief Title: Comparison Study of Usual Care vs. Usual Care Plus Community Intervention to Manage Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Ontario Ministry of Health and Long Term Care (Other Government); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Maureen Markle-Reid, RN, PhD, Scientific Director, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: DRCT-06669
Record Dates: First submitted 2014-06-03; First posted 2014-06-09 (Estimated); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: Type 2 Diabetes Mellitus; NIDDM; Non-insulin Dependent Diabetes Mellitus
Keywords: Self-Management; Home Visits
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — House Calls

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Primary Care (No Intervention): Usual Primary Care will be received by half the participants during the course of the Study
- Home Visits and educational support (Active Comparator): Intervention comprised of Home Visits and group educational sessions. Home Visits and will be conducted by Diabetes Education staff in lieu of usual care conducted at the Diabetes clinic. Lifestyle support and educational will be offered in the form of monthly Diabetes Wellness Days offered in the community where nutrition, exercise and support will be given to help improve self-management of diabetes.
  Interventions: Behavioral: Home Visits and Lifestyle Education Support

INTERVENTIONS:
Behavioral: Home Visits and Lifestyle Education Support
  Arms: Home Visits and educational support

SUMMARY:
The overall purpose of this research is to examine and compare the effectiveness and costs of a community-based intervention to support self-management with usual primary care for older adults with Type 2 Diabetes Mellitus and multiple chronic conditions and their family caregivers. Once the study is complete, the investigators will be able to determine if there is any measurable difference in self-care management between usual care plus the intervention versus usual care alone.

DETAILED DESCRIPTION:
Research Goal

To examine the comparative effectiveness and costs of a community-based intervention to support self-management with usual primary care for older adults with T2DM and Multiple Chronic Conditions and their family caregivers.

Objectives

1. To determine if a 6-month, IP, community-based intervention improve self-management compared with usual primary care services?
2. To compare the effectiveness of the intervention on HRQoL, physical activity, nutritional status, depression, anxiety, diabetes parameters (blood glucose levels [HbA1c, hypoglycemic episodes]), diabetes-related complications, number of vascular events, social support number of falls, fall risk and medication safety with usual primary care services?
3. To determine the effectiveness of the intervention on HRQoL of family caregivers compared with usual primary care?
4. To assess whether or not the intervention improves clinical practice behaviours?
5. To determine the 6-month costs of use of health services of the intervention compared with usual care, from a social perspective?
6. To identify which subgroups of older adults with T2DM and MCC benefit most from the intervention?
7. To determine the effectiveness of the intervention based on sex/gender and region?
8. To determine the overall feasibility and acceptability of an IP community-based health promotion intervention and what can be identified as barriers and facilitators to implementation?

ELIGIBILITY:
Inclusion Criteria:

* older adults aged 65+
* live in the local vicinity of a participating Diabetes Education Program
* were referred to their Diabetes Education Program within the past 24 months
* competence in English (or access to a translator)
* intention to continue living in the area for the next 6 months
* two reported chronic conditions in addition to T2DM. Individuals with newly diagnosed T2DM as well as those who were already receiving treatment for T2DM will be eligible for inclusion in the study.

Exclusion Criteria:

* score of 20 or less in Montreal Cognitive Assessment (MoCA) test AND without access to a substitute decision maker to sign consent (Score of 20 or less is not in itself an exclusion).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 291 (Actual)
Dates: Start 2014-09; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Summary of Diabetes Self-Care Activities | Every two months from study onset until the end of study (6 months from baseline)
  The SDSCA is a multidimensional measure of diabetes self-management with adequate internal and test-retest reliability, and evidence of validity and sensitivity to change. The revised SDSCA consists of items that assess the following aspects of the diabetes regimen: general and specific diet, exercise, blood-glucose testing, foot care, and smoking. Scores are calculated for each of these five regimen areas. This data is collected by the interventionists at each visit.

SECONDARY OUTCOMES:
SF12v2 | Baseline and end of study (6 months from baseline)
  This measurement is used to assess Health related quality of Life. This survey consists of 12 questions that measure functional health and well-being from the client's perspective. It provides scores for eight health domains (physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, mental health), and psychometrically-based physical component summary (PCS) and mental component summary (MCS) scores

OTHER OUTCOMES:
CES-D-10 | Baseline and end of study (6 months from baseline)
  The CES-D has been used in prior studies of older adults with mood disorders, and has a high degree of reliability, content, construct and criterion related validity, distinguishes between depressed and non-depressed people, and is a sensitive tool for measuring changes in depressive symptoms over time in psychiatric populations.
GAD-7 | Baseline and end of study (6 months from baseline)
  Prevalence and severity of anxiety, measured by the Generalized Anxiety Disorder Screener
Health Assessment forms | Baseline intervention interview, at 3 months and again at 6 months
  • Diabetes parameters (fasting blood glucose, HbA1c, hypoglycemic episodes), and presence of diabetes-related complications and comorbid chronic conditions, obtained from health assessment forms submitted by the Diabetes Education Program RN and RD after the first home visit and at 3 months and 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Maureen Markle-Reid, PhD, Principal Investigator — McMaster University; Jenny Ploeg, PhD, Principal Investigator — McMaster University
Locations (8):
- Canada (8):
  - Edmonton Oliver PCN, Edmonton, Alberta
  - Leduc Beaumont Devon PCN, Leduc, Alberta
  - Sherwood Park PCN, Sherwood Park, Alberta
  - McMaster University, Hamilton, Ontario
  - Ross Memorial Hospital, Lindsay, Ontario
  - St. Joseph's Health Care, London, Ontario
  - Peterborough Regional Health Centre, Peterborough, Ontario
  - Port Hope Community Health Centre, Port Hope, Ontario

REFERENCES:
- [Result] Markle-Reid M, Ploeg J, Fraser KD, Fisher KA, Bartholomew A, Griffith LE, Miklavcic J, Gafni A, Thabane L, Upshur R. Community Program Improves Quality of Life and Self-Management in Older Adults with Diabetes Mellitus and Comorbidity. J Am Geriatr Soc. 2018 Feb;66(2):263-273. doi: 10.1111/jgs.15173. Epub 2017 Nov 27. PMID 29178317
- [Derived] Miklavcic JJ, Fraser KD, Ploeg J, Markle-Reid M, Fisher K, Gafni A, Griffith LE, Hirst S, Sadowski CA, Thabane L, Triscott JAC, Upshur R. Effectiveness of a community program for older adults with type 2 diabetes and multimorbidity: a pragmatic randomized controlled trial. BMC Geriatr. 2020 May 13;20(1):174. doi: 10.1186/s12877-020-01557-0. PMID 32404059
- [Derived] Markle-Reid M, Ploeg J, Valaitis R, Duggleby W, Fisher K, Fraser K, Ganann R, Griffith LE, Gruneir A, McAiney C, Williams A. Protocol for a program of research from the Aging, Community and Health Research Unit: Promoting optimal aging at home for older adults with multimorbidity. J Comorb. 2018 Jul 31;8(1):2235042X18789508. doi: 10.1177/2235042X18789508. eCollection 2018. PMID 30191144
- [Derived] Markle-Reid M, Ploeg J, Fraser KD, Fisher KA, Akhtar-Danesh N, Bartholomew A, Gafni A, Gruneir A, Hirst SP, Kaasalainen S, Stradiotto CK, Miklavcic J, Rojas-Fernandez C, Sadowski CA, Thabane L, Triscott JA, Upshur R. The ACHRU-CPP versus usual care for older adults with type-2 diabetes and multiple chronic conditions and their family caregivers: study protocol for a randomized controlled trial. Trials. 2017 Feb 6;18(1):55. doi: 10.1186/s13063-017-1795-9. PMID 28166816